CLINICAL TRIAL: NCT04586413
Title: Post Acute COVID-19 Quality of Life (PAC-19QoL) Tool Development and Patient Registry (PAC-19QoLReg)
Status: Recruiting | Type: Observational
Sponsor: Medialis Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Med_Asst 33
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Covid19
Keywords: Covid19; Quality of Life; Post-Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-hospitalised post-COVID-19 patients: This cohort will have had a confirmed positive test for COVID-19 or antibody test confirming they had COVID-19 but they were not hospitalised for this
  Interventions: Other: No intervention - quality of life measure
- Hospitalised post-COVID-19 patients: This cohort will have a confirmed diagnosis of COVID-19 and been hospitalised but were not in an Intensive Care Unit
  Interventions: Other: No intervention - quality of life measure
- Intensive care post-COVID-19 patients: This cohort will have a confirmed diagnosis of COVID-19 and been hospitalised in an Intensive Care Unit
  Interventions: Other: No intervention - quality of life measure

INTERVENTIONS:
Other: No intervention - quality of life measure — Participants will be part of the creation of a Post-COVID-19 quality of life measure if involved in Phase One. In Phase Two participants will complete this post-COVID-19 quality of life measure monthly for 12 months

SUMMARY:
Coronavirus Disease 2019 (COVID-19) is a newly emerged disease, caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The COVID-19 pandemic is having a large impact on the mental and physical health of patients, yet data on the quality of life of post-COVID-19 patients is lacking. There are currently no post-COVID-19 specific measures for quality of life, particularly none which include the views of post-COVID-19 patients themselves. This observational study will recruit participants to contribute their preferences to the creation of a post-COVID-19 specific patient-reported measure on post-COVID-19 quality of life. Participants will be split into three groups: those who were not hospitalised; those who were hospitalised but not in intensive care units; and those who were hospitalised and in intensive care units. The creation of this measure will form phase 1 of the study, with 30-60 participants (10-20 in each group above) recruited to complete online surveys to find out their preferences of areas of life to include in such a measure. This will involve 3 online surveys, 1) to ask which areas of life they feel are impacted and how; 2) to find consensus about the areas to be included; 3) to weight the relevance of these areas in relation to each other. In phase 2 recruitment will open to additional participants and all participants will be asked to complete the finalised post-COVID-19 quality of life measure once a month for 12 months, aiming for a minimum of 100 participants at this stage. All participants will also be asked to complete a demographic questionnaire to inform the analysis of the data.

DETAILED DESCRIPTION:
This observational study will be conducted in two phases:

Phase 1 - the development of a post-COVID-19 patient reported quality of life measure Phase 2 - the longitudinal completion of the quality of life tool by post-COVID-19 patients each month for 12 months All participants will complete an online informed consent form and a demographic questionnaire at the start of their involvement with the study Phase 1 The study will recruit a minimum of 30 participants and a maximum of 60 participants, 10-20 across three groups: those who were not hospitalised; those who were hospitalised but not in intensive care units; and those who were hospitalised and in intensive care units. Investigators will take the first 10-20 participants who match in each group. If contact is received from participants but their group is already full they will be asked if they are still be happy to participate in phase 2 and an offer to contact them when that commences will be made.

Firstly, a novel method (Jandhyala Method) will be used to elicit post-COVID-19 patients' preferences for a post-COVID-19 quality of life tool. Participants will do this by completing an Awareness Round survey, this means using free-text responses to ask participants about the areas of their lives impacted by COVID-19 and those areas they see as most important to their quality of life. The research team will collate and code these free text responses then create a comprehensive list of all of those deemed important to participants who will then be sent a Consensus Round survey to ask how far they agree or disagree with the inclusion of those items in a quality of life tool. Researchers will then collate this information, group it into relevant domains and develop a weighting tool to be sent to participants to ask them to rate the relevant importance of the different areas to be included, which will be used to create weighted domain and item scores to be used in a final quality of life tool. We expect for the Awareness round surveys to be completed within a one month time period and then two weeks will be allocated for the research team to analyse and finalise the Consensus round survey; the Consensus round survey will then be open for two weeks, with prompting to participants after one week if not completed. The research team will then have a further two weeks to complete the weighting tool and participants will be given a further two weeks to complete this. At this stage the research team will have a further two weeks to finalise the Post-COVID-19 quality of life tool and then phase 2 will begin.

In summary:

1. Awareness round online survey (hosted on Survey Monkey) - asking for areas of life which the participants feel have been impacted by COVID-19, including details and examples of those impacts

   a. The research team will collate and code these responses and generate a list of statements based on the information provided by participants
2. Consensus round online survey (hosted on Survey Monkey) - the list of statements will be sent to participants and they will be asked to rate how far they agree or disagree with the inclusion of these areas in a post-COVID-19 quality of life tool

   a. The research team will collate this information, group it into relevant domains and develop a weighting tool
3. Weighting tool (online Microsoft excel template) - participants will be asked to weight the individual items and domains for the finalised post-COVID-19 quality of life tool using an online excel spreadsheet template a. The research team will use this information to develop the finalised post-COVID-19 quality of life measure to be completed by participants and to develop the system to score this tool Phase 2 At this stage the recruitment will be re-opened for additional participants, including those with a clinical diagnosis regardless of test status, aiming for a minimum of 100 and a maximum of 5000 at this stage, though this will be subject to review. Recruitment will remain open for time 1 surveys for one year, with a another year following this to gain the full 12 months of data from participants, again subject to review. The finalised post-COVID-19 quality of life measure will be hosted on a secure online system (Castor EDC tm) and participants will be allocated an ID number. They will be asked to complete this measure at monthly intervals for a period of 12 months. The research team will analyse the changes over time within and between groups. Statistical methods for this will be finalised when the measure has been completed at the end of Phase 1 by our biostatistician.

ELIGIBILITY:
Phase One

Inclusion Criteria:

* The participant has had either a confirmed COVID-19 test while infected or a confirmed COVID-19 antibody test post-infection
* The participant is aged 18 years or older
* The participant is capable of providing informed consent
* The participant can read, write and converse in English
* The participant can comply with the study schedule

Exclusion Criteria:

* The participant does not have a confirmed COVID-19 test or antibody test
* The participant is aged under 18 years
* The participant is not capable of giving informed consent
* The participant is unable to read, write and converse in English
* The participant is unable to comply with study schedule data collection

Phase Two

Inclusion Criteria:

* The participant has had either a confirmed COVID-19 test while infected or a confirmed COVID-19 antibody test post-infection or a clinical diagnosis of COVID-19
* The participant is aged 18 years or older
* The participant is capable of providing informed consent
* The participant can read, write and converse in English
* The participant can comply with the study schedule

Exclusion Criteria:

* The participant does not have a confirmed COVID-19 test or antibody test or clinical diagnosis of COVID-19
* The participant is aged under 18 years
* The participant is not capable of giving informed consent
* The participant is unable to read, write and converse in English
* The participant is unable to comply with study schedule data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have a confirmed diagnosis of COVID-19 from either a test while infected or an antibody test post infection for Phase One. Participants in Phase Two will have either confirmed test/antibody test or clinical diagnosis of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Design of PAC19QoL Measure (Phase One) | 3 months
  The design and creation of a Post-COVID-19 Quality of Life Measure
Completion of PAC19QoL Measure monthly for 12 months (Phase Two) | 12 months
  Participants in Phase Two will complete the newly designed Post-COVID-19 quality of life measure each month for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Jandhyala, Study Chair — Medialis Ltd.
Locations (1):
- Medialis, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD

REFERENCES:
- [Derived] Jandhyala R. Design, validation and implementation of the post-acute (long) COVID-19 quality of life (PAC-19QoL) instrument. Health Qual Life Outcomes. 2021 Sep 28;19(1):229. doi: 10.1186/s12955-021-01862-1. PMID 34583690
- See also: Publication — https://pubmed.ncbi.nlm.nih.gov/37675987/
- See also: Related Info — https://hqlo.biomedcentral.com/articles/10.1186/s12955-021-01862-1#:~:text=The%20PAC%2D19QoL%20instrument%20for,affected%20their%20quality%20of%20life.